CLINICAL TRIAL: NCT02424851
Title: A Study of Thalidomide, Bendamustine and Dexamethasone (BTD) Versus Bortezomib, Bendamustine and Dexamethasone (BBD) in Patients With Renal Failure Defined as a GFR Below 30 Mls/Min
Brief Title: Optimising Renal Outcome in Myeloma Renal Failure
Acronym: OPTIMAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: Janssen-Cilag Ltd. (Industry); Bloodwise (Other); University of Warwick (Other); University of Birmingham (Other)
Responsible Party: Principal Investigator, Karthik Ramasamy, Dr., Oxford University Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26866138-MMY2070; 2012-003947-31 (EudraCT Number)
Record Dates: First submitted 2015-03-10; First posted 2015-04-23 (Estimated); Results first posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Multiple Myeloma; Chronic Kidney Disease
Keywords: myeloma; multiple myeloma; chronic kidney disease; renal failure; bortezomib; Velcade; thalidomide; bendamustine; dexamethasone; serum free light chains; proteosomal inhibition; immunomodulatory
MeSH Terms: conditions — Multiple Myeloma; Renal Insufficiency, Chronic; Neoplasms, Plasma Cell; Renal Insufficiency | interventions — Bortezomib; Thalidomide; Bendamustine Hydrochloride; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (BBD) (Active Comparator): Bortezomib, Bendamustine and Dexamethasone
  Interventions: Drug: Bortezomib; Drug: Bendamustine; Drug: Dexamethasone
- Arm B (BTD) (Active Comparator): Thalidomide, Bendamustine and Dexamethasone
  Interventions: Drug: Thalidomide; Drug: Bendamustine; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bortezomib — 1.3 mg/m2 subcutaneously* days 1, 4, 8 and 11 of each cycle. Number of cycles: Four 21 day cycles (participants not suitable for ASCT (autologous stem cell transplant) will continue up to 6 cycles on the treatment regimen to which they were randomised).
  *intravenous infusion available in case of patient intolerance to subcutaneous bortezomib
  Other Names: Velcade
  Arms: Arm A (BBD)
Drug: Thalidomide — 100 mg daily orally, preferably at night, days 1-21 of each cycle. Four 21 day cycles (participants not suitable for ASCT will continue up to 6 cycles on the treatment regimen to which they were randomised)
  Arms: Arm B (BTD)
Drug: Bendamustine — 60 mg/m2 i.v. days 1 and 8 of each cycle. Four 21 day cycles (participants not suitable for ASCT will continue up to 6 cycles on the treatment regimen to which they were randomised)
Drug: Dexamethasone — 40mg orally days 1-2, 4-5, 8-9 and 11-12 of each cycle

SUMMARY:
The purpose of this study is to compare the effectiveness of bortezomib versus thalidomide in reducing free light chains in the blood of myeloma patients. In addition participants will receive bendamustine (chemotherapy) and dexamethasone (steroids), which increase the effectiveness of both bortezomib and thalidomide. The trial will also study whether an earlier reduction of free light chains increases the chances of the kidneys recovering.

DETAILED DESCRIPTION:
Renal impairment is a life threatening condition of myeloma. 20-25% of patients will present at diagnosis with renal dysfunction. Outcome is poor due to high early mortality, with 28% of newly diagnosed myeloma patients in myeloma trials with renal failure not surviving beyond 100 days, compared with 10% overall.

This study aims to establish:

1. Whether proteosomal inhibition (bortezomib) or immunomodulatory (thalidomide) based therapy achieves threshold reduction of serum free light chains (sFLCs) in a significant majority of patients.
2. Whether sFLC response to the first 2 cycles (early responder) predicts haematological and renal response to the next 2 cycles of therapy.
3. An early time point for assessment of sFLC reduction as a biomarker for response.

Participants will be stratified by age and chronic kidney disease (CKD) stage to receive either bortezomib, bendamustine and dexamethasone (BBD) or thalidomide, bendamustine and dexamethasone (BTD).

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial.
* Patients attending NHS (National Health Service) Haemato-oncology centres.
* Patients with newly diagnosed symptomatic myeloma.
* Glomerular Filtration Rate (GFR) <30 mls/min.
* Chronic kidney disease (CKD) staging is based on estimated or measured GFR. CKD stage 4 (15-29 ml/min) and CKD stage 5 (<15 ml/min) are eligible to enter the study. It is expected centres will consider use of fluid resuscitation and pulsed dose of steroid therapy in this group of patients to salvage renal function prior to trial screening.
* A number of patients with newly diagnosed myeloma and renal failure will have a pre-existing medical condition (hypertension, diabetes etc.) causing renal damage. Where there is a medical condition (e.g. hypertension, diabetes) which may cause renal damage, there must have been a further decline (≥15 mls/min GFR) between previous steady state and the study screening.
* Female participants of childbearing potential and male patients whose partner is a woman of childbearing potential must be prepared to use contraception in accordance with (and consent to) the Celgene-approved process for thalidomide and lenalidomide Risk Management and Pregnancy Prevention Programme.
* Women of childbearing potential must have a negative pregnancy test performed by a healthcare professional in accordance with the Celgene-approved process for thalidomide and lenalidomide Risk Management and Pregnancy Prevention.
* Free of prior malignancies for ≥ 2 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, localised prostate cancer or carcinoma "in-situ" of the cervix or breast.
* In the Investigator's opinion, is able and willing to comply with all trial requirements.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the trial.

Exclusion Criteria:

* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial or the female partner of a male participant planning a pregnancy during the course of the trial.
* Known allergy to investigational drugs.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Any of the following laboratory abnormalities:
* Absolute neutrophil count (ANC) < 1.0 x10^9/L
* Platelet count <75 x 10^9/L
* Serum SGOT/AST or SGPT/ALT (serum glutamic oxaloacetic transaminase/aspartate aminotransferase or serum glutamic pyruvic transaminase/alanine aminotransferase) >3 x upper limit of normal.
* Use of any standard/experimental anti-myeloma drug therapy excluding dexamethasone 14 days prior to trial entry.
* CKD stages < 4.
* Intention to use a physical method of serum free light chain removal such as plasma exchange or high cut off dialysis.
* Grade 2 neuropathy or more (National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v 4.0) will preclude use of thalidomide and bortezomib.
* Participants who have participated in another research trial involving an investigational product in the past 12 weeks.
* Contraindicated to receive either one of the study drugs, thalidomide, bortezomib, bendamustine based on the respective summary of product characteristics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-11; Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karthik Ramasamy, Principal Investigator — National Health Service, United Kingdom
Locations (9):
- United Kingdom (9):
  - Basingstoke & North Hampshire Hospital, Basingstoke
  - Heartlands Hospitals, Birmingham
  - Kent & Canterbury Hospital, Canterbury
  - St Helier Hospital, Epsom
  - Royal Liverpool Hospital, Liverpool
  - Kings College Hospital, London
  - Churchill Hospital, Oxford
  - Queen Alexandra Hospital, Portsmouth
  - Great Western Hospital, Swindon

REFERENCES:
- [Background] Kumar SK, Rajkumar SV, Dispenzieri A, Lacy MQ, Hayman SR, Buadi FK, Zeldenrust SR, Dingli D, Russell SJ, Lust JA, Greipp PR, Kyle RA, Gertz MA. Improved survival in multiple myeloma and the impact of novel therapies. Blood. 2008 Mar 1;111(5):2516-20. doi: 10.1182/blood-2007-10-116129. Epub 2007 Nov 1. PMID 17975015
- [Background] Brenner H, Gondos A, Pulte D. Expected long-term survival of patients diagnosed with multiple myeloma in 2006-2010. Haematologica. 2009 Feb;94(2):270-5. doi: 10.3324/haematol.13782. Epub 2009 Jan 14. PMID 19144659
- [Background] Landgren O, Kyle RA, Pfeiffer RM, Katzmann JA, Caporaso NE, Hayes RB, Dispenzieri A, Kumar S, Clark RJ, Baris D, Hoover R, Rajkumar SV. Monoclonal gammopathy of undetermined significance (MGUS) consistently precedes multiple myeloma: a prospective study. Blood. 2009 May 28;113(22):5412-7. doi: 10.1182/blood-2008-12-194241. Epub 2009 Jan 29. PMID 19179464
- [Background] Knudsen LM, Hippe E, Hjorth M, Holmberg E, Westin J. Renal function in newly diagnosed multiple myeloma--a demographic study of 1353 patients. The Nordic Myeloma Study Group. Eur J Haematol. 1994 Oct;53(4):207-12. doi: 10.1111/j.1600-0609.1994.tb00190.x. PMID 7957804
- [Background] Eleutherakis-Papaiakovou V, Bamias A, Gika D, Simeonidis A, Pouli A, Anagnostopoulos A, Michali E, Economopoulos T, Zervas K, Dimopoulos MA; Greek Myeloma Study Group. Renal failure in multiple myeloma: incidence, correlations, and prognostic significance. Leuk Lymphoma. 2007 Feb;48(2):337-41. doi: 10.1080/10428190601126602. PMID 17325894
- [Background] Clark AD, Shetty A, Soutar R. Renal failure and multiple myeloma: pathogenesis and treatment of renal failure and management of underlying myeloma. Blood Rev. 1999 Jun;13(2):79-90. doi: 10.1016/s0268-960x(99)90014-0. PMID 10414944
- [Background] Drayson M, Begum G, Basu S, Makkuni S, Dunn J, Barth N, Child JA. Effects of paraprotein heavy and light chain types and free light chain load on survival in myeloma: an analysis of patients receiving conventional-dose chemotherapy in Medical Research Council UK multiple myeloma trials. Blood. 2006 Sep 15;108(6):2013-9. doi: 10.1182/blood-2006-03-008953. Epub 2006 May 25. PMID 16728700
- [Background] Morgan GJ, Davies FE, Gregory WM, Bell SE, Szubert AJ, Navarro Coy N, Cook G, Feyler S, Johnson PR, Rudin C, Drayson MT, Owen RG, Ross FM, Russell NH, Jackson GH, Child JA; National Cancer Research Institute Haematological Oncology Clinical Studies Group. Cyclophosphamide, thalidomide, and dexamethasone as induction therapy for newly diagnosed multiple myeloma patients destined for autologous stem-cell transplantation: MRC Myeloma IX randomized trial results. Haematologica. 2012 Mar;97(3):442-50. doi: 10.3324/haematol.2011.043372. Epub 2011 Nov 4. PMID 22058209
- [Background] Augustson BM, Begum G, Dunn JA, Barth NJ, Davies F, Morgan G, Behrens J, Smith A, Child JA, Drayson MT. Early mortality after diagnosis of multiple myeloma: analysis of patients entered onto the United kingdom Medical Research Council trials between 1980 and 2002--Medical Research Council Adult Leukaemia Working Party. J Clin Oncol. 2005 Dec 20;23(36):9219-26. doi: 10.1200/JCO.2005.03.2086. Epub 2005 Nov 7. PMID 16275935
- [Background] Torra R, Blade J, Cases A, Lopez-Pedret J, Montserrat E, Rozman C, Revert L. Patients with multiple myeloma requiring long-term dialysis: presenting features, response to therapy, and outcome in a series of 20 cases. Br J Haematol. 1995 Dec;91(4):854-9. doi: 10.1111/j.1365-2141.1995.tb05400.x. PMID 8547129
- [Background] Kastritis E, Anagnostopoulos A, Roussou M, Gika D, Matsouka C, Barmparousi D, Grapsa I, Psimenou E, Bamias A, Dimopoulos MA. Reversibility of renal failure in newly diagnosed multiple myeloma patients treated with high dose dexamethasone-containing regimens and the impact of novel agents. Haematologica. 2007 Apr;92(4):546-9. doi: 10.3324/haematol.10759. PMID 17488666
- [Background] Knudsen LM, Hjorth M, Hippe E. Renal failure in multiple myeloma: reversibility and impact on the prognosis. Nordic Myeloma Study Group. Eur J Haematol. 2000 Sep;65(3):175-81. doi: 10.1034/j.1600-0609.2000.90221.x. PMID 11007053
- [Background] Alexanian R, Barlogie B, Dixon D. Renal failure in multiple myeloma. Pathogenesis and prognostic implications. Arch Intern Med. 1990 Aug;150(8):1693-5. PMID 2383164
- [Background] Gandhi V. Metabolism and mechanisms of action of bendamustine: rationales for combination therapies. Semin Oncol. 2002 Aug;29(4 Suppl 13):4-11. doi: 10.1053/sonc.2002.34872. PMID 12170425
- [Background] Gaul L, Mandl-Weber S, Baumann P, Emmerich B, Schmidmaier R. Bendamustine induces G2 cell cycle arrest and apoptosis in myeloma cells: the role of ATM-Chk2-Cdc25A and ATM-p53-p21-pathways. J Cancer Res Clin Oncol. 2008 Feb;134(2):245-53. doi: 10.1007/s00432-007-0278-x. Epub 2007 Jul 25. PMID 17653574
- [Background] Ponisch W, Mitrou PS, Merkle K, Herold M, Assmann M, Wilhelm G, Dachselt K, Richter P, Schirmer V, Schulze A, Subert R, Harksel B, Grobe N, Stelzer E, Schulze M, Bittrich A, Freund M, Pasold R, Friedrich T, Helbig W, Niederwieser D; East German Study Group of Hematology and Oncology (OSHO). Treatment of bendamustine and prednisone in patients with newly diagnosed multiple myeloma results in superior complete response rate, prolonged time to treatment failure and improved quality of life compared to treatment with melphalan and prednisone--a randomized phase III study of the East German Study Group of Hematology and Oncology (OSHO). J Cancer Res Clin Oncol. 2006 Apr;132(4):205-12. doi: 10.1007/s00432-005-0074-4. Epub 2006 Jan 10. PMID 16402269
- [Background] Knop S, Straka C, Haen M, Schwedes R, Hebart H, Einsele H. The efficacy and toxicity of bendamustine in recurrent multiple myeloma after high-dose chemotherapy. Haematologica. 2005 Sep;90(9):1287-8. PMID 16154860
- [Background] Haubitz M, Bohnenstengel F, Brunkhorst R, Schwab M, Hofmann U, Busse D. Cyclophosphamide pharmacokinetics and dose requirements in patients with renal insufficiency. Kidney Int. 2002 Apr;61(4):1495-501. doi: 10.1046/j.1523-1755.2002.00279.x. PMID 11918757
- [Background] Eriksson T, Hoglund P, Turesson I, Waage A, Don BR, Vu J, Scheffler M, Kaysen GA. Pharmacokinetics of thalidomide in patients with impaired renal function and while on and off dialysis. J Pharm Pharmacol. 2003 Dec;55(12):1701-6. doi: 10.1211/0022357022241. PMID 14738599
- [Background] Tosi P, Zamagni E, Cellini C, Cangini D, Tacchetti P, Tura S, Baccarani M, Cavo M. Thalidomide alone or in combination with dexamethasone in patients with advanced, relapsed or refractory multiple myeloma and renal failure. Eur J Haematol. 2004 Aug;73(2):98-103. doi: 10.1111/j.1600-0609.2004.00272.x. PMID 15245508
- [Background] Morgan GJ, Davies FE, Gregory WM, Russell NH, Bell SE, Szubert AJ, Navarro Coy N, Cook G, Feyler S, Byrne JL, Roddie H, Rudin C, Drayson MT, Owen RG, Ross FM, Jackson GH, Child JA; NCRI Haematological Oncology Study Group. Cyclophosphamide, thalidomide, and dexamethasone (CTD) as initial therapy for patients with multiple myeloma unsuitable for autologous transplantation. Blood. 2011 Aug 4;118(5):1231-8. doi: 10.1182/blood-2011-02-338665. Epub 2011 Jun 7. PMID 21652683
- [Background] Ramasamy K, Hazel B, Mahmood S, Corderoy S, Schey S. Bendamustine in combination with thalidomide and dexamethasone is an effective therapy for myeloma patients with end stage renal disease. Br J Haematol. 2011 Dec;155(5):632-4. doi: 10.1111/j.1365-2141.2011.08754.x. Epub 2011 Jun 21. No abstract available. PMID 21689088
- [Background] Jagannath S, Barlogie B, Berenson JR, Singhal S, Alexanian R, Srkalovic G, Orlowski RZ, Richardson PG, Anderson J, Nix D, Esseltine DL, Anderson KC; SUMMIT/CREST Investigators. Bortezomib in recurrent and/or refractory multiple myeloma. Initial clinical experience in patients with impared renal function. Cancer. 2005 Mar 15;103(6):1195-200. doi: 10.1002/cncr.20888. PMID 15690325
- [Background] Chanan-Khan AA, Kaufman JL, Mehta J, Richardson PG, Miller KC, Lonial S, Munshi NC, Schlossman R, Tariman J, Singhal S. Activity and safety of bortezomib in multiple myeloma patients with advanced renal failure: a multicenter retrospective study. Blood. 2007 Mar 15;109(6):2604-6. doi: 10.1182/blood-2006-09-046409. Epub 2006 Nov 30. PMID 17138816
- [Background] San Miguel JF, Schlag R, Khuageva NK, Dimopoulos MA, Shpilberg O, Kropff M, Spicka I, Petrucci MT, Palumbo A, Samoilova OS, Dmoszynska A, Abdulkadyrov KM, Schots R, Jiang B, Mateos MV, Anderson KC, Esseltine DL, Liu K, Cakana A, van de Velde H, Richardson PG; VISTA Trial Investigators. Bortezomib plus melphalan and prednisone for initial treatment of multiple myeloma. N Engl J Med. 2008 Aug 28;359(9):906-17. doi: 10.1056/NEJMoa0801479. PMID 18753647
- [Background] Fenk R, Michael M, Zohren F, Graef T, Czibere A, Bruns I, Neumann F, Fenk B, Haas R, Kobbe G. Escalation therapy with bortezomib, dexamethasone and bendamustine for patients with relapsed or refractory multiple myeloma. Leuk Lymphoma. 2007 Dec;48(12):2345-51. doi: 10.1080/10428190701694194. PMID 18067009
- See also: Cancer Research UK - Myeloma Statistics — http://www.cancerresearchuk.org/cancer-info/cancerstats/types/myeloma/uk-multiple-myeloma-statistics

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (BBD): Bortezomib, Bendamustine and Dexamethasone
  Bortezomib: 1.3 mg/m2 subcutaneously* days 1, 4, 8 and 11 of each cycle. Number of cycles: Four 21 day cycles (participants not suitable for ASCT (autologous stem cell transplant) will continue up to 6 cycles on the treatment regimen to which they were randomised).
  *intravenous infusion available in case of patient intolerance to subcutaneous bortezomib
  Bendamustine: 60 mg/m2 i.v. days 1 and 8 of each cycle. Four 21 day cycles (participants not suitable for ASCT will continue up to 6 cycles on the treatment regimen to which they were randomised)
  Dexamethasone: 40mg orally days 1-2, 4-5, 8-9 and 11-12 of each cycle
Period: Overall Study
Arm/Group | Arm A (BBD) | Arm B (BTD)
Started | 16 | 15
Completed | 14 | 12
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (BBD) | Arm B (BTD) | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Customized [Count of Participants; unit: Participants]
  ≤70 years | 8 | 8 | 16
  >70 years | 8 | 7 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 8 | 9 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 16 | 15 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With >50% Reduction From Baseline in Serum Free Light Chain
Time Frame: End of week 6 (after receiving two cycles of therapy)
Population: The primary endpoint of serum free light chain response was assessed in 30 patients where samples were available at screening and the end of two cycles of trial treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (BBD) | Arm B (BTD)
Number analyzed (Participants) | 16 | 14
Participants | 13 | 3
Statistical Analysis 1: Comparison: Arm A (BBD) vs Arm B (BTD); Test type: Other; p = 0.006, Fisher Exact

2. Primary Outcome: Number of Participants With Different Renal Responses to Treatment
Time Frame: End of week 12 (after receiving 4 cycles of therapy)
Population: Renal response in accordance with IMWG criteria was assessed in 20 patients with eGFR and creatinine clearance data recorded at screening and at the end of four cycles of trial treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (BBD) | Arm B (BTD)
Number analyzed (Participants) | 16 | 15
Participants
  Complete/partial response | 5 | 1
  Minor response | 3 | 7
  No response | 3 | 1
  Not evaluable | 5 | 6
Statistical Analysis 1: Comparison: Arm A (BBD) vs Arm B (BTD); Test type: Other; p = 0.02, Fisher Exact

3. Secondary Outcome: Haematological and Non-haematological Toxicity in Both Treatment Arms
Time Frame: End of weeks 3, 6, 9, 12 (after receiving 4 cycles of therapy), 30 days after final treatment and 12 months after randomisation
Measure: Number; unit: Events
Arm/Group | Arm A (BBD) | Arm B (BTD)
Number analyzed (Participants) | 16 | 15
Events
  Serious adverse events | 2 | 0
  Adverse events | 3 | 6
Statistical Analysis 1: Comparison: Arm A (BBD) vs Arm B (BTD); Statistical analysis of SAEs; Test type: Other; p = 0.48, Fisher Exact
Statistical Analysis 2: Comparison: Arm A (BBD) vs Arm B (BTD); Statistical analysis of AEs; Test type: Other; p = 0.25, Fisher Exact

4. Secondary Outcome: Overall Survival
Time Frame: 1 month post end of treatment and 1 year post randomisation
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (BBD) | Arm B (BTD)
Number analyzed (Participants) | 16 | 15
Participants | 9 | 13
Statistical Analysis 1: Comparison: Arm A (BBD) vs Arm B (BTD); Test type: Other; p = 0.31, Log Rank

5. Secondary Outcome: Renal Response After Two Cycles of Trial Treatment
Time Frame: End of 2nd treatment cycle, week 6
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (BBD) | Arm B (BTD)
Number analyzed (Participants) | 15 | 13
Participants
  Partial response | 2 | 0
  Minor response | 9 | 7
  No repsonse | 4 | 6
Statistical Analysis 1: Comparison: Arm A (BBD) vs Arm B (BTD); Test type: Other; p = 0.45, Fisher Exact

6. Secondary Outcome: Quality of Life Measured by the EQ-5D-3L Questionnaire at Baseline and 1 Month Follow up
Description: The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension is scored on a scale of 1 to 3: 1 (no problems), 2 (some problems), and 3 (extreme problems). Higher score equates to a worse outcome.
  As stated in the official EQ-5D user guide, patient responses to the 5 questions were converted into a single index value as per Dolan P (1997). Modeling valuations for EuroQol health states. Med Care 35(11):1095-108. These index values, with country specific value sets, facilitate the calculation of quality-adjusted life years (QALYs) that are used to inform economic evaluations of health care interventions. In the UK, the values range from -0.594 to +1.
Time Frame: Baseline and 1 month follow up
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Arm A (BBD) | Arm B (BTD)
Number analyzed (Participants) | 8 | 9
Units on a scale
  Baseline | 0.72 (0.15) | 0.69 (0.35)
  1 month FU | 0.69 (0.19) | 0.80 (0.28)
Statistical Analysis 1: Comparison: Arm A (BBD) vs Arm B (BTD); Test type: Other; p = 0.33, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 4 years, 2 months.
Arm/Group | Arm A (BBD) | Arm B (BTD)
All-Cause Mortality (participants affected / at risk) | 7/16 | 2/15
Serious Adverse Events (participants affected / at risk) | 11/16 | 9/15
Other Adverse Events (participants affected / at risk) | 15/16 | 11/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (BBD) (N=16) | Arm B (BTD) (N=15)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bone infection (Infections and infestations) | 1 (1) | 0 — Osteomyelitis
Bronchial infection (Infections and infestations) | 1 (2) | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 2 (2)
Delirium (Psychiatric disorders) | 0 | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 | 1 (1)
Edema limbs (General disorders) | 1 (1) | 0
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0
Fatigue (General disorders) | 0 | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 (1)
Fever (General disorders) | 0 | 2 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Hematuria (Renal and urinary disorders) | 0 | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 0 | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 0
Skin infection (Infections and infestations) | 1 (1) | 0 — Cellulitis
Stroke (Nervous system disorders) | 0 | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0
Thromboembolic event (Vascular disorders) | 0 | 1 (1) — PE
Transient ischemic attacks (Nervous system disorders) | 1 (1) | 0
Upper respiratory infection (Infections and infestations) | 2 (2) | 0
Urinary tract infection (Infections and infestations) | 0 | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (BBD) (N=16) | Arm B (BTD) (N=15)
Alanine aminotransferase increased (Investigations) | 0 | 1 (1)
Alkaline Phosphatase Increased (Investigations) | 0 | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (4)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0
Anxiety (Psychiatric disorders) | 1 (1) | 0
Bone infection (Infections and infestations) | 1 (1) | 0
Bronchial Infection (Infections and infestations) | 1 (1) | 0
Catheter related infection (Infections and infestations) | 1 (1) | 0
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fever (General disorders) | 1 (1) | 1 (1)
Weight Loss (Investigations) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 3 (4)
Tremor (Nervous system disorders) | 1 (1) | 3 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (8)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Conjunctivtis (Eye disorders) | 1 (1) | 0
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0
Insomnia (Psychiatric disorders) | 1 (1) | 0
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Mucosal infection (Infections and infestations) | 1 (1) | 0
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify: Labial cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0
Papulopustular rash (Infections and infestations) | 1 (1) | 0
Blurred vision (Eye disorders) | 1 (2) | 0
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (2) | 0
Syncope (Nervous system disorders) | 1 (2) | 0
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Skin infection (Infections and infestations) | 2 (2) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 2 (5)
Paresthesia (Nervous system disorders) | 2 (2) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (3) | 2 (2)
Edema limbs (General disorders) | 4 (4) | 3 (3)
Fatigue (General disorders) | 4 (4) | 5 (9)
Lung infection (Infections and infestations) | 2 (5) | 3 (5)
Nausea (Gastrointestinal disorders) | 4 (5) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (6) | 2 (3)
Constipation (Gastrointestinal disorders) | 4 (11) | 3 (3)
Chronic Kidney Disease (Renal and urinary disorders) | 0 | 1 (1)
Creatinine increased (Investigations) | 0 | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 | 1 (1)
Eye disorders - Other, specify: visual disturbance? (Eye disorders) | 0 | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 (1)
Hypertension (Vascular disorders) | 0 | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 (1)
Hypotension (Vascular disorders) | 0 | 1 (1)
Infections and infestations - Other, specify: infection (unknown source) (Infections and infestations) | 0 | 1 (1)
Infusion Site Extravasation (General disorders) | 0 | 1 (1)
Left Ventricular systolic dysfunction (Cardiac disorders) | 0 | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
Oral Dysesthesia (Gastrointestinal disorders) | 0 | 1 (1)
Pain (General disorders) | 0 | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
Presyncope (Nervous system disorders) | 0 | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)
Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 1 (1)
Superficial thrombophlebitis (Vascular disorders) | 0 | 1 (1)
Thromboembolic event (Vascular disorders) | 0 | 1 (1)
Erythroderma (Skin and subcutaneous tissue disorders) | 0 | 1 (2)
Palmar-plantae erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 (2)
Infections and infestations - Other, specify: (Oral) thrush (Infections and infestations) | 0 | 2 (2)
Lymphocyte count decreased (Investigations) | 0 | 2 (2)
Stomach pain (Gastrointestinal disorders) | 0 | 2 (2)
White blood cell decreased (Investigations) | 0 | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT02424851/Prot_SAP_000.pdf